CLINICAL TRIAL: NCT04604158
Title: IIT2020-13-GRESHAM-ELLY: Evaluating the Effect of a Mobile Audio Companion (Elly) to Reduce Anxiety in Cancer Patients
Brief Title: Evaluating the Effect of a Mobile Audio Companion (Elly) to Reduce Anxiety in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gillian Gresham (Other)
Responsible Party: Sponsor-Investigator, Gillian Gresham, Principal Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2020-13-GRESHAM-ELLY
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Cancer Metastatic; Neoplasms; Breast Cancer; Lung Cancer; Glioblastoma; Prostate Cancer; Gynecologic Cancer; Colorectal Cancer; Sarcoma; Kidney Cancer; Bladder Cancer; Lymphoma; Leukemia; Head and Neck Cancer; Pancreas Cancer; Multiple Myeloma; Anxiety; Social Isolation; Stress; Loneliness; Melanoma; Uterine Cancer
Keywords: Elly Health; Elly App
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Breast Neoplasms; Lung Neoplasms; Glioblastoma; Prostatic Neoplasms; Colorectal Neoplasms; Sarcoma; Kidney Neoplasms; Urinary Bladder Neoplasms; Lymphoma; Leukemia; Head and Neck Neoplasms; Pancreatic Neoplasms; Multiple Myeloma; Anxiety Disorders; Social Isolation; Melanoma; Uterine Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elly Mobile Phone Application (Experimental)
  Interventions: Behavioral: Elly Mobile Phone Application

INTERVENTIONS:
Behavioral: Elly Mobile Phone Application — The Elly mobile phone application delivers daily audio recording aimed at reducing anxiety, stress, loneliness, and social isolation.
  Other Names: Elly App

SUMMARY:
This is a single-arm, prospective, interventional study in cancer survivors and patients to examine the feasibility of a mobile health application, Elly (Elly Health Inc.), to reduce levels of anxiety, stress, loneliness, and social isolation. Participants will be given access to the Elly phone application developed by Elly Health Inc. and will be asked to complete questionnaires measuring quality of life at multiple timepoints during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer of any type and currently receiving cancer-targeted treatment or have received cancer-targeted treatment within 6 months of consent date based on self-report. Cancer-targeted treatment includes chemotherapy, radiation therapy, hormonal therapy, biologic therapy, immunotherapy, and surgery.
* 18 years or older
* Access to and ability to use an iPhone (SE+, iOS 12.4+)
* Ability to understand and read English
* Have an understanding, ability, and willingness to fully comply with study procedures and restrictions

Exclusion Criteria:

- Hearing loss or vision impairment that would preclude the participant from accessing and using the app (use of hearing aids or visual aids is acceptable) based on self-report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Absolute change in patient-reported anxiety scores at Day 30 compared with baseline. | 30 days
  Absolute change in patient-reported anxiety scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 30 compared with baseline. The minimum value is 6 and maximum value is 30, and a lower score means a better outcome.

SECONDARY OUTCOMES:
Absolute change in patient-reported anxiety scores at Day 14 compared with baseline. | 14 days
  Absolute change in patient-reported anxiety scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 14 compared with baseline. The minimum value is 6 and maximum value is 30, and a lower score means a better outcome.
Absolute change in patient-reported anxiety scores at Day 60 compared with baseline. | 60 days
  Absolute change in patient-reported anxiety scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 60 compared with baseline. The minimum value is 6 and maximum value is 30, and a lower score means a better outcome.
Absolute change in patient-reported anxiety scores at Day 90 compared with baseline. | 90 days
  Absolute change in patient-reported anxiety scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 90 compared with baseline. The minimum value is 6 and maximum value is 30, and a lower score means a better outcome.
Absolute change in patient-reported anxiety scores at Day 120 compared with baseline. | 120 days
  Absolute change in patient-reported anxiety scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 120 compared with baseline. The minimum value is 6 and maximum value is 30, and a lower score means a better outcome.
Absolute change in patient-reported anxiety scores at Day 150 compared with baseline. | 150 days
  Absolute change in patient-reported anxiety scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 150 compared with baseline. The minimum value is 6 and maximum value is 30, and a lower score means a better outcome.
Absolute change in patient-reported anxiety scores at Day 180 compared with baseline. | 180 days
  Absolute change in patient-reported anxiety scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 180 compared with baseline. The minimum value is 6 and maximum value is 30, and a lower score means a better outcome.
Absolute change in patient-reported depression scores at Day 30 compared with baseline. | 30 days
  Absolute change in patient-reported depression scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 30 compared with baseline. The minimum value is 8 and maximum value is 40, and a lower score means a better outcome.
Absolute change in patient-reported depression scores at Day 60 compared with baseline. | 60 days
  Absolute change in patient-reported depression scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 60 compared with baseline. The minimum value is 8 and maximum value is 40, and a lower score means a better outcome.
Absolute change in patient-reported depression scores at Day 90 compared with baseline. | 90 days
  Absolute change in patient-reported depression scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 90 compared with baseline. The minimum value is 8 and maximum value is 40, and a lower score means a better outcome.
Absolute change in patient-reported depression scores at Day 120 compared with baseline. | 120 days
  Absolute change in patient-reported depression scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 120 compared with baseline. The minimum value is 8 and maximum value is 40, and a lower score means a better outcome.
Absolute change in patient-reported depression scores at Day 150 compared with baseline. | 150 days
  Absolute change in patient-reported depression scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 150 compared with baseline. The minimum value is 8 and maximum value is 40, and a lower score means a better outcome.
Absolute change in patient-reported depression scores at Day 180 compared with baseline. | 180 days
  Absolute change in patient-reported depression scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 180 compared with baseline. The minimum value is 8 and maximum value is 40, and a lower score means a better outcome.
Absolute change in patient-reported loneliness scores at Day 30 compared with baseline. | 30 days
  Absolute change in patient-reported loneliness scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 30 compared with baseline. The minimum value is 5 and maximum value is 25, and a lower score means a better outcome.
Absolute change in patient-reported loneliness scores at Day 60 compared with baseline. | 60 days
  Absolute change in patient-reported loneliness scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 60 compared with baseline. The minimum value is 5 and maximum value is 25, and a lower score means a better outcome.
Absolute change in patient-reported loneliness scores at Day 90 compared with baseline. | 90 days
  Absolute change in patient-reported loneliness scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 90 compared with baseline. The minimum value is 5 and maximum value is 25, and a lower score means a better outcome.
Absolute change in patient-reported loneliness scores at Day 120 compared with baseline. | 120 days
  Absolute change in patient-reported loneliness scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 120 compared with baseline. The minimum value is 5 and maximum value is 25, and a lower score means a better outcome.
Absolute change in patient-reported loneliness scores at Day 150 compared with baseline. | 150 days
  Absolute change in patient-reported loneliness scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 150 compared with baseline. The minimum value is 5 and maximum value is 25, and a lower score means a better outcome.
Absolute change in patient-reported loneliness scores at Day 180 compared with baseline. | 180 days
  Absolute change in patient-reported loneliness scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 180 compared with baseline. The minimum value is 5 and maximum value is 25, and a lower score means a better outcome.
Absolute change in patient-reported social isolation scores at Day 30 compared with baseline. | 30 days
  Absolute change in patient-reported social isolation scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 30 compared with baseline. The minimum value is 4 and maximum value is 20, and a lower score means a better outcome.
Absolute change in patient-reported social isolation scores at Day 60 compared with baseline. | 60 days
  Absolute change in patient-reported social isolation scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 60 compared with baseline. The minimum value is 4 and maximum value is 20, and a lower score means a better outcome.
Absolute change in patient-reported social isolation scores at Day 90 compared with baseline. | 90 days
  Absolute change in patient-reported social isolation scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 90 compared with baseline. The minimum value is 4 and maximum value is 20, and a lower score means a better outcome.
Absolute change in patient-reported social isolation scores at Day 120 compared with baseline. | 120 days
  Absolute change in patient-reported social isolation scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 120 compared with baseline. The minimum value is 4 and maximum value is 20, and a lower score means a better outcome.
Absolute change in patient-reported social isolation scores at Day 150 compared with baseline. | 150 days
  Absolute change in patient-reported social isolation scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 150 compared with baseline. The minimum value is 4 and maximum value is 20, and a lower score means a better outcome.
Absolute change in patient-reported social isolation scores at Day 180 compared with baseline. | 180 days
  Absolute change in patient-reported social isolation scores as measures using the NIH (National Institutes of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire at Day 180 compared with baseline. The minimum value is 4 and maximum value is 20, and a lower score means a better outcome.
Frequency of Elly app use | 180 days
  Frequency of study participant opening the Elly app
Elly app login amount (frequency and duration) | 180 days
  Number of logins to Elly app by study participant
Feasibility | 180 days
  Download of Elly app and engage with app at least 40% 3 or more times over study period.
Participant's experience with Elly app at Day 14-30. | Day 30
  Participant's experience with Elly app based on qualitative interview done between Day 14-30.
Participant's experience with Elly app at Day 180-360. | Day 360
  Participant's experience with Elly app based on qualitative interview done between Day 180-360.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Gresham, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No